CLINICAL TRIAL: NCT06817031
Title: Ability of the Probiotic VE818 to Reduce Enteropathogen Colonization and Improve Environmental Enteropathy in Pregnant Women: A Proof-of-Concept and Phase II Randomized Placebo-Controlled Trial in Bangladesh, Pakistan, Zambia, and Burkina Faso
Brief Title: Maternal Probiotic Intervention to Improve Gut Health - Trial II - Bangladesh
Acronym: MPIGH-II
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-24002
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Environmental Enteric Dysfunction
Keywords: probiotic, environmental enteropathy, pregnancy, maternal, gut health, microbiome
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observation only arm (No Intervention)
- oral vancomycin + placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Oral Vancomycin
- oral vancomycin + VE818 (Active Comparator)
  Interventions: Drug: VE818; Drug: Oral Vancomycin

INTERVENTIONS:
Drug: VE818 — VE818, is an 11-strain bacterial consortium rationally designed by Vedanta Biosciences Inc., to displace enteropathogens and reduce intestinal inflammation in pregnant women
  Arms: oral vancomycin + VE818
Drug: Placebo — Enteric Capsules filled with approximately 400mg of Microcrystalline Cellulose (bulking agent)
  Arms: oral vancomycin + placebo
Drug: Oral Vancomycin — Oral vancomycin in capsule form will be administered three times daily for 5 days at 250mg per dose. Because oral vancomycin is a non-absorbable antibiotic, the likelihood of systemic absorption is minimal and therefore, it is not associated with the adverse events attributable to the intravenous formulation
  Arms: oral vancomycin + VE818; oral vancomycin + placebo

SUMMARY:
Burden: Environmental Enteric Dysfunction (EED) is an enteropathic condition characterised by altered gut permeability, infiltration of immune cells and changes in villous architecture and cell differentiation. EED is a major reason of malnourishment, poor neurological development, stunting, oral vaccine failure, and infection. It is believed that EED is responsible for 40% of all childhood stunting.

Knowledge gap: To date the focus of research on childhood stunting has been on the young child. It is increasingly appreciated, however, that stunting often begins in utero and the focus has shifted to women's health and pregnancy. Results from rural Bangladesh reveal poor gestational weight gain that ultimately leads to intrauterine growth restriction, low birth weight and ultimately stunting and wasting. Another study recently completed in slum settlements of Dhaka, Bangladesh demonstrated a high prevalence of EED among undernourished women. Intestinal histopathology was abnormal in more than 80% of women. We postulate that growth retardation in utero is a consequence of EED in the mother during pregnancy and lactation. This leads to systemic inflammation, which lead to disadvantageous partitioning of nutrients, and reduced nutrient availability.

Relevance: This trial will explore the conceptual framework that a probiotic or live biotherapeutic product that can improve the composition of gut microbiota, can also displace enteropathogens and reduce biomarkers of intestinal inflammation to promote gut health. This will restore healthy microbial signalling to the host epithelium, ameliorate barrier function through secretion of mucus and antimicrobial factors, and improve nutrient availability.

Objectives: The primary objective is to assess if administration of oral vancomycin followed by VE818 to pregnant women colonised with at least 2 out of 11 selected bacterial enteropathogens results in a significant change in the mean count of these organisms between the baseline and 2 weeks after completion of the intervention (Study Day 35d +2), compared to oral vancomycin followed by placebo.

Methods: Pregnant women will be recruited in antenatal clinics and in the community in Matlab in Bangladesh, Matiari in Pakistan, Lusaka in Zambia and, and Bobo-Dioulasso in Burkina Faso. Study population will be women aged 18 years or older in the first trimester or early second trimester of pregnancy. Study procedures will be explained in detail and written consent will be taken before enrollment. Those women who give consent to participation will undergo a screening process which will check if any exclusion criteria are fulfilled. After consent and screening they will be randomised into either of the three arms: intervention arm (oral vancomycin followed by VE818), placebo-control arm (oral vancomycin followed by placebo), or observation-only arm. The allocation sequence will be generated by the trial statistician using a code with block permutation. The participant will remain free to withdraw at any time from the trial without giving reasons and without prejudicing her further treatment. Biological samples, including blood, saliva, urine, stool, vaginal swab, and intestinal luminal contents through CapScan. CapScan is a non-invasive device (capsule) that collects gastrointestinal samples along the gastrointestinal tract following ingestion and passes into stool.

Outcome measures/variables: The primary endpoint is the change in the mean count in the number of 11 selected fecal bacterial pathogen groups present between baseline and 2 weeks after completion of the 14-day course with Placebo or VE818 (Study arms 2 and 3), which corresponds to 35th day, +2 from the first dose of oral vancomycin.

The 11 enteropathogen targets will be detected by customized real-time quantitative PCR-based TaqMan Array Cards (TAC-qPCR) and include the following organisms: Aeromonas, Campylobacter coli, Campylobacter jejuni, Campylobacter Pan, Enteroaggregative Escherichia coli (E. coli), Enteropathogenic E. coli, Enterotoxigenic E. coli, Plesiomonas, Shigella_Enteroinvasive E. coli (EIEC), Salmonella and Klebsiella pneumoniae

DETAILED DESCRIPTION:
Across the site pregnant women will be screened for eligibility in their first or early second trimester of pregnancy (13-17 weeks of GA) and will be enrolled and randomized into three arms (48 women per arm). Participants will be dosed depending on the randomized arm.

As per WHO recommendation, participants in all 3 arms will receive Multiple Micronutrient Supplements (MMS) as part of routine antenatal care, which they will begin taking at enrollment and continue throughout pregnancy.

Blinding will be implemented for the comparison between the Treatment arm and the Placebo arm. However, it is not feasible to apply blinding to the Observation-only arm as the participants in this group will receive no intervention and the arm solely serves as an observational arm.

After the end of the intervention, pregnant women will be followed up until birth to record birth and pregnancy outcomes. Mother-infant dyads will be sampled 7 days after birth. Maternal and Infant health outcomes will be followed up to 1 month after childbirth to record clinical outcomes during this period.

ELIGIBILITY:
All pregnant women in their first or early second trimester of pregnancy, residing in the icddr,b service area of Matlab, who meet the eligibility criteria decribed below.

Inclusion criteria

1. Women aged 18 years or older in their first or early second trimester of pregnancy (13-17 weeks of gestational age [GA]), living in defined geographical areas of Bangladesh (Matlab), Pakistan, Zambia, and Burkina Faso, where it can be assumed that environmental enteropathy is prevalent

   AND
2. Presence of any 2 out of 11 selected bacterial pathogen targets (Aeromonas, Campylobacter coli, Campylobacter jejuni, Campylobacter Pan, Enteroaggregative Escherichia coli, Enteropathogenic Escherichia coli, Enterotoxigenic Escherichia coli, Plesiomonas, Shigella_EIEC, Salmonella and Klebsiella pneumoniae in fecal samples measured by TAC-qPCR.

   AND
3. Presence of any of the following WASH conditions -

   1. use surface water, unimproved water, or limited water for drinking; OR
   2. use surface water, unimproved water, or limited water for cooking; OR
   3. use surface water, unimproved water, or limited water for washing utensils; OR
   4. practice open defecation, use unimproved sanitation (toilet facility), or limited sanitation (toilet facility); OR
   5. lack facility or have limited facility for handwashing

Exclusion criteria

Potential participants will not be enrolled if they:

1. have MUAC ≥30 cm
2. are carrying more than one fetus (i.e., multiple pregnancy)
3. have diarrhea, defined as the passage of three or more loose stools per 24 hours, or have had diarrhea in the preceding 14 days
4. have fever or an active infection
5. have taken antibiotics or probiotics in the preceding 14 days
6. have taken steroids or non-steroidal anti-inflammatory drugs in the preceding 14 days
7. have severe anemia as determined using finger stick Hb < 8 g/dl
8. have a history of chronic digestive disease
9. have any gastrointestinal contraindication to ingestion of a capsule (known or suspected gastrointestinal obstruction, stricture, fistula, gastroparesis, or any swallowing disorder)
10. have known immunocompromised status (known history of HIV infection, autoimmune disease, diabetes mellitus, etc.)
11. have known drug hypersensitivity/allergy/intolerance
12. have chronic disease or any other illness or condition which in the opinion of the investigator will complicate the assessment of safety or efficacy
13. are medically disqualified: Any potential participant who is deemed medically unfit for trial enrollment by a non-study healthcare provider, due to the presence of severe or unstable health conditions that could compromise safety or interfere with the study outcomes, will be excluded from participation
14. have a plan to observe fast any time during the intervention period
15. have a plan to leave the study area within the follow-up period
16. are participating in any other interventional trial
17. belong to a household from which another woman is already enrolled in the study

but may be enrolled if/when these disqualifiers have expired.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in the mean count in the number of 11 selected fecal bacterial pathogen groups present between baseline and endline | Between baseline and 2 weeks after completion of the 14-day course with Placebo or VE818
  The primary endpoint is the change in the mean count in the number of 11 selected fecal bacterial pathogen groups present between baseline and 2 weeks after completion of the 14-day course with Placebo or VE818 (Study arms 2 and 3), which corresponds to 35th day, +2 from the first dose of oral vancomycin.

SECONDARY OUTCOMES:
Change in prevalence of specific enteropathogens not included in the primary endpoint in pregnant women | Baseline, day 6, day 21, day 35, day 63 and 7 day post-partum
  Change in prevalence of specific enteropathogens (i.e., rotavirus, norovirus, Giardia, Cryptosporidium, and bacterial pathogens not included in the primary endpoint) in pregnant women detected in feces by TAC-qPCR between baseline (Day 0), end of oral vancomycin treatment (Day 6) the last dose of the 14-day VE818 intervention (21st day, +2), 14 days after the last dose of VE818 (35th day, +2), 42 days after the last dose of VE818 (63rd day, +2), and 7 day post-partum in the Treatment arm compared to Placebo arm and Observation-only arm (comparable timepoints)
Engraftment of VE818 strains in pregnant women | day 21, day 35, day 63 and 7 day post-partum
  Engraftment of VE818 strains in pregnant women as measured by shotgun metagenomic sequencing of fecal samples collected at the end of the 14-day VE818 intervention (21st day, +2), 14 days after the last dose of VE818 (35th day, +2), 42 days after the last dose of VE818 (63rd day, +2) and 7 days post-partum
Change in a panel of plasma biomarkers in pregnant women as measured by ELISA | Baseline, day 6, day 35, and day 63
  Change in a panel of plasma biomarkers (CRP, AGP, sCD14, LBP, CD163 and iFABP) in pregnant women as measured by ELISA between baseline (Day 0), end of oral vancomycin treatment (Day 6), 14 days after the last dose the of 14-day intervention (35th day, +2) and, 42 days after the last dose of VE818 (63rd day, +2) in the Treatment arm compared to Placebo arm and Observation-only arm (comparable timepoints)
Change in a panel of fecal biomarkers in pregnant women as measured by ELISA | Baseline, day 6, day 21, day 35, day 63 and 7 day post-partum
  Change in a panel of fecal biomarkers (myeloperoxidase, neopterin, calprotectin and lipocalin) in pregnant women as measured by ELISA between baseline (Day 0) , end of oral vancomycin treatment (Day 6), the last dose of the 14-day VE818 intervention (21st day, +2), 14 days after the last dose of VE818 (35th day, +2) 42 days after the last dose VE818 (63rd day, +2), and 7 day post-partum in the Treatment arm, compared to Placebo arm and Observation-only arm (comparable timepoints)
Change in intestinal permeability as measured by Lactulose/Rhamnose (LR) ratio in pregnant women | Baseline and day 35
  Change in intestinal permeability as measured by Lactulose/Rhamnose (LR) ratio in pregnant women between baseline and 14 days after the last dose of 14-day VE818 intervention (35th day, +2) in the Treatment arm, compared to Placebo arm and Observation-only arm (comparable timepoints)
Change in alpha and beta diversity of fecal microbiome in pregnant women | Baseline, day 6, day 21, day 35, day 63 and 7 day post-partum
  Change in alpha and beta diversity of fecal microbiome in pregnant women as measured by shotgun metagenomics sequencing between baseline (Day 0), end of oral vancomycin treatment (Day 6), the last dose of the 14-day VE818 intervention (21st day, +2), 14 days after the last dose of VE818 (35th day, +2 day), 42 days after the last dose of VE818 (63rd day, +2), and 7 day post-partum in the Treatment arm, compared to Placebo arm and Observation-only arm ( comparable timepoints)
Change in alpha and beta diversity of vaginal microbiome in pregnant women | Baseline, day 6, day 35, and day 63
  Change in alpha and beta diversity of vaginal microbiome in pregnant women as measured by shotgun metagenomics sequencing between baseline, end of oral vancomycin treatment (Day 6), 14 days after the last dose of the 14-day VE818 intervention (35th day, +2), and 42 days after the last dose of VE818 (63rd day, +2), in the Treatment arm, compared to Placebo arm and Observation-only arm (comparable timepoints)
Change in alpha and beta diversity of oral microbiome in pregnant women | Baseline and day 35
  Change in alpha and beta diversity of oral microbiome in pregnant women as measured by shotgun metagenomics sequencing between baseline (Day 0) (and 14 days after the last dose of the 14-day VE818 intervention (35th day, +2), in the Treatment arm, compared to Placebo arm and Observation-only arm (comparable timepoints)
Change in metabolome (plasma and stool) in pregnant women | Baseline, day 6, day 21, day 35, day 63 and 7 day post-partum
  Change in metabolome (plasma, and stool) in pregnant women between baseline (Day 0), end of oral vancomycin treatment (Day 6), the last dose of the 14-day VE818 intervention (21st day +2; stool only), 14 days after the last dose of VE818 (35th day+2) 42 days after the last dose of VE818 (63rd day +2) and 7 days post birth (stool only) in the Treatment arm, compared to Placebo arm and Observation-only arm (comparable timepoints)

OTHER OUTCOMES:
Difference in the rate of weight gain during the second and third trimester of pregnancy | Second and third trimester of pregnancy
  Difference in the rate of weight gain during the second and third trimester of pregnancy between Treatment arm and Placebo and Observation-only arms
Difference in fetal growth trajectories | 16 weeks, 20 weeks, 24 weeks, 28 weeks, 32 weeks and 36 weeks of gestation
  Difference in fetal growth trajectories as measured by serial ultrasound evaluation of intrauterine growth between Treatment arm and Placebo and Observation-only arms
Difference in placental insufficiency | 28 weeks, 32 weeks, and 36 weeks of gestation
  Difference in placental insufficiency as measured by ultrasound-derived cerebroplacental ratio (CPR) between Treatment arm and Placebo and Observation-only arms
Difference in placental stress | First, second, and third trimester of pregnancy
  Difference in placental stress measured through sFlt-1/PlGF ratio between Treatment arm and Placebo and Observation-only arms
Change in alpha and beta diversity in the gut microbiota of pregnant women | Baseline and day 35
  Change in alpha and beta diversity in the gut microbiota of pregnant women as measured by shotgun metagenomic sequencing of intestinal fluid obtained using CapScan between baseline and 14 days after the last dose of the 14-day VE818 intervention (35th day, +2), in the Treatment arm, compared to Placebo arm and Observation-only arm (comparable timepoints)
Engraftment of VE818 strains in CapScan samples | Baseline and day 35
  Engraftment of VE818 strains in CapScan samples collected 14 days after the last dose of VE818 (35th day, +2) as measured by shotgun metagenomic sequencing
Difference in average count of enteropathogens in infants | 7 days post birth
  Difference in average count of enteropathogens in infants detected in feces by TAC-qPCR 7 days after birth between Treatment arm and Placebo and Observation-only arms
Difference in a panel of fecal biomarkers in infants | 7 days post birth
  Difference in a panel of fecal biomarkers (myeloperoxidase, neopterin, calprotectin and lipocalin) in infants as measured by ELISA 7 days after birth between Treatment arm and Placebo and Observation-only arms
Difference in alpha and beta diversity of fecal microbiome in infants | 7 days post birth
  Difference in alpha and beta diversity of fecal microbiome in infants as measured by shotgun metagenomics sequencing 7 days after birth between Treatment arm and Placebo and Observation-only arms
Detection of VE818 organisms in infants | 7 days post birth
  Detection of VE818 organisms in infants measured via metagenomic analysis of fecal samples collected 7 days after birth
Difference in fecal metabolome in infants | 7 days post birth
  Difference in fecal metabolome in infants 7 days after birth between Treatment arm, Placebo arm and Observation-only arms
Variability in endpoint assays across geographies and laboratories | Baseline, day 6, day 21, day 35, day 63 and 7 day post-partum
  Variability in endpoint assays across geographies and laboratories
Difference in perinatal outcomes | Perinatal period
  Difference in perinatal outcomes between Treatment arm, Placebo arm and Observation-only arms
Difference in birth anthropometry | At birth
  Difference in birth anthropometry between Treatment arm, Placebo arm and Observation-only arms
Difference in growth measures and morbidity of the infants | 1 month post birth
  Differences in growth measures and morbidity of the infants 1 month post birth between Treatment arm, Placebo arm and Observation-only arms
Difference in women's postpartum weight change | 1 month post-partum
  Differences in women's postpartum weight change (loss/retention) between Treatment arm, Placebo arm and Observation-only arms
Difference in maternal immune responses | Baseline, day 6, day 35, day 63, and 7 days and 1 month post-partum
  Differences in maternal immune responses in plasma, cord blood and breast milk between Treatment arm, Placebo arm and Observation-only arms (comparable timepoints)
Difference in gene expression in maternal and infant stool samples | Baseline, day 6, day 21, day 35, day 63 and 7 days post birth
  Differences in gene expression in maternal and infant stool samples between Treatment arm, Placebo arm and Observation-only arms (comparable timepoints)

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Chāndpur, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided